CLINICAL TRIAL: NCT05939089
Title: Cardiovascular Assessment of Pediatric Cancer Survivors: Understanding Long-Term Effects and Risks
Brief Title: Cardiovascular Assessment of Pediatric Cancer Survivors
Acronym: CASPER
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cafer Zorkun, Head, Division of CardioOncology, Istanbul University
Other Study IDs: COEXIST-2
Record Dates: First submitted 2023-06-24; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Left Ventricular Dysfunction; Heart Failure
Keywords: Childhood Cancer Survivors; Cardiotoxicity; cancer treatment related heart diseases
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure; Cardiotoxicity | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG, Echocardiography, cTnI, NT-ProBNP — All pediatric cancer survivors are evaluated with cardiological examination, ECG, transthoracic echocardiography (transesophageal echocardiography when required), NT-proBNP, cTnI, kidney function tests, liver function tests, fasting blood glucose, cholesterol panel, iron, iron binding capacity, ferritin, transferrin saturation, B12, vitamin D, folic acid, urinanalysis, hemogram and a questionnaire about living with heart failure.

SUMMARY:
The goal of this observational study is to evaluate cardiac and vascular health status of pediatric cancer survivors.

DETAILED DESCRIPTION:
All pediatric cancer survivors were evaluated with cardiological examination, ECG, transthoracic echocardiography (transesophageal echocardiography when required), NT-proBNP, cTnI, kidney function tests, liver function tests, fasting blood glucose, cholesterol panel, iron, iron binding capacity, ferritin, transferrin saturation, B12, vitamin D, folic acid, urinanalysis, hemogram and a questionnaire about living with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cancer at pediatric age

Exclusion Criteria:

* Having cancer after 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are less than 18 years-old, diagnosed and treated for any type of cancer.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Rate of LV Dysfunction | From the first visit at cardio-oncology division through study completion, an average of 2 years
  Echocardiographic evaluation of left ventricular functions

CONTACTS AND LOCATIONS:
Overall Officials: Cafer Zorkun, MD PhD, Principal Investigator — Faculty member
Locations (1):
- Istanbul Faculty of Medicine, Fatih, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing study data in a public place, requires additional (written) permission from all participants, and then from local IRB.